CLINICAL TRIAL: NCT04544956
Title: B-Fine: An Open Label, Single Arm Study to Mechanistically Interrogate the Therapeutic Effect of GSK3228836 in Patients With Chronic Hepatitis B Via Intrahepatic Immunophenotyping
Brief Title: A Mechanistic Study of GSK3228836 With Fine Needle Aspiration (FNA) in Participants With Chronic Hepatitis B
Acronym: B-Fine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 212602
Record Dates: First submitted 2020-09-04; First posted 2020-09-10 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-04

CONDITIONS: Hepatitis B
Keywords: Hepatitis B virus; GSK3228836; Fine needle aspiration; Intrahepatic immunophenotyping
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Intervention Model Description: A single arm, multi-center, open label exploratory study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GSK3228836 300 mg (Experimental): Participants on stable nucleos(t)ide therapy will receive GSK3228836 300 mg subcutaneously (SC) weekly once for 12 weeks along with a loading dose of GSK3228836 300 mg in Week 1 (Day 4) and Week 2 (Day 11).
  Interventions: Drug: GSK3228836; Drug: Nucleos(t)ide therapy

INTERVENTIONS:
Drug: GSK3228836 — GSK3228836 will be available as a clear colorless to slightly yellow solution for injection in 150 mg/milliliters (mL) vial to be administered SC once weekly.
Drug: Nucleos(t)ide therapy — Participants receiving nucleos(t)ide therapy upon entry in the study will continue to receive nucleos(t)ide therapy for the duration of the study.

SUMMARY:
Hepatitis B virus (HBV) infection, especially chronic, is a significant worldwide medical problem. This is an exploratory study of the therapeutic mechanism of GSK3228836 in participants with chronic hepatitis B (CHB) on stable nucleos(t)ide therapy (which is the first line therapy for CHB). This study is a Phase IIa, multi-center open label exploratory study of the therapeutic mechanism of GSK3228836 in participants with hepatitis B virus e-antigen (HBeAg)-negative CHB on stable nucleos(t)ide therapy using repeat fine needle aspirations of the liver for intrahepatic immunophenotyping. It will investigate the virologic and immunologic correlates of hepatitis B virus surface antigen (HBsAg) loss observed in participants when treated for 12 weeks with 300 milligrams (mg) GSK3228836. Repeat fine needle aspirates of the liver will be performed to enable analysis of liver-resident immune cells to investigate any immunomodulatory properties of GSK3228836 and to study the biology of underlying treatment-associated liver flares. The study will consist of a screening, treatment, and post-treatment follow-up phase. Approximately 20 participants will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be at least 18 years of age at the time of signing the informed consent.
* Participants who have documented chronic HBV infection >=6 months prior to screening and currently receiving stable nucleos(t)ide analogue therapy, defined as no changes to their nucleos(t)ide regimen from at least 6 months prior to screening and with no planned changes to the stable regimen over the duration of the study.
* Plasma or serum HBsAg concentration >100 IU/mL
* Plasma or serum HBV DNA concentration must be adequately suppressed, defined as plasma or serum HBV DNA <90 IU/mL.
* HBeAg-negative
* ALT less than or equal to (<=)2 times ULN
* No gender restriction.
* A male participant is eligible to participate if they agree to the following during the intervention period and for at least 90 days after the last dose of study treatment i. Refrain from donating sperm ii. and be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or Must agree to use contraception/barrier as detailed below

  1) Agree to use a male condom (and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak) when having sexual intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant.
* A female participant is eligible to participate:

  i. If she is not pregnant or breastfeeding. ii. and at least one of the following conditions applies:
  1. Is not a WOCBP
  2. or is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1 percent [%] per year), preferably with low user dependency during the intervention period and for at least 90 days after the last dose of study treatment iii. A WOCBP must have both

  <!-- -->

  1. A confirmed menstrual period prior to the first dose of study intervention (additional evaluation [e.g. amenorrhea in athletes, birth control] should also be considered)
  2. and a negative highly sensitive pregnancy test (urine or serum) within 24 hours before the first dose of study treatment
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Clinically significant abnormalities, aside from chronic HBV infection in medical history (e.g., moderate-severe liver disease other than chronic HBV, acute coronary syndrome within 6 months of screening, major surgery within 3 months of screening, significant/unstable cardiac disease, uncontrolled diabetes, bleeding diathesis or coagulopathy) or physical examination.
* Co-infection with:

  1. Current or past history of Hepatitis C virus (HCV)
  2. Human immunodeficiency virus (HIV)
  3. Hepatitis D virus (HDV).
* History of or suspected liver cirrhosis and/or evidence of cirrhosis as determined by

  1. Both Aspartate aminotransferase (AST)-Platelet Index (APRI) >2 and FibroSure/FibroTest result >0.7

     1) If only one parameter (APRI or FibroSure/FibroTest) result is positive, a discussion with the Medical Monitor is required before inclusion in study is permitted.
  2. Regardless of APRI or Fibrosure/FibroTest score participants will be excluded from the study if their past history includes one of the following criteria:

     1. Liver biopsy showing Metavir 4 or equivalent
     2. Liver stiffness >12 kilopascals (kPa)
* Diagnosed or suspected hepatocellular carcinoma as evidenced by the following

  1. Alpha-fetoprotein concentration >=200 nanograms (ng)/mL
  2. If the screening alpha fetoprotein concentration is >=50 ng/mL and <200 ng/mL, the absence of liver mass must be documented by imaging within 6 months before enrolment.
* History of malignancy within the past 5 years with the exception of specific cancers that are cured by surgical resection (e.g., skin cancer). Participants under evaluation for possible malignancy are not eligible.
* History of vasculitis or presence of symptoms and signs of potential vasculitis (e.g., vasculitic rash, skin ulceration, repeated blood detected in urine without identified cause) or history/presence of other diseases that may be associated with vasculitis condition (e.g., systemic lupus erythematosus, rheumatoid arthritis, relapsing polychondritis, mononeuritis multiplex).
* History of extrahepatic disorders possibly related to HBV immune conditions (e.g., nephrotic syndrome, any type of glomerulonephritis, polyarteritis nodosa, cryoglobulinemia, uncontrolled hypertension).
* Anti-neutrophil cytoplasmic antibody (ANCA) at screening by itself won't be an exclusion criterion - but if results are borderline positive or positive:

  1. Myeloperoxidase (MPO)-ANCA (perinuclear [p] ANCA) and Proteinase 3 (PR3)-ANCA (Cytoplasmic [c] ANCA) analysis will be conducted
  2. A discussion with the Medical Monitor will be required to review participant's complete medical history to ensure no past history or current manifestations of a vasculitic/inflammatory/auto-immune condition before inclusion in study is permitted.
* Low compliment (C)3 at screening or Baseline by itself won't be an exclusion criterion-but if it is present

  a. A discussion with the Medical Monitor is required to review participant's complete medical history to ensure no past history or current manifestations of vasculitic/inflammatory/auto-immune conditions.
* History of alcohol or drug abuse/dependence

  1. Current alcohol use as judged by investigator to potentially interfere with participant compliance.
  2. History of or current drug abuse/dependence as judged by the investigator to potentially interfere with participant compliance.

     1. Refers to illicit drugs and substances with abuse potential. Medications that are used by the participant as directed, whether over-the-counter or through prescription, are acceptable and would not meet the exclusion criteria.
* Currently taking, or took within 3 months of screening, any immunosuppressing drugs (e.g., prednisone), other than a short course of therapy (<=2 weeks) or topical/inhaled steroid use.
* Participants for whom immunosuppressive treatment is not advised, including therapeutic doses of steroids, will be excluded.
* Currently taking, or took within 12 months of screening, any interferon-containing therapy.
* Participants requiring anti-coagulation therapies (for example warfarin, Factor Xa inhibitors or anti-platelet agents like clopidogrel).
* The participant has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 5 half-lives (if known) or twice the duration (if known) of the biological effect of the study treatment (whichever is longer) or 90 days (if half-life or duration is unknown).
* Prior treatment with any oligonucleotide or small interfering RNA (siRNA) within 12 months prior to the first dosing day.
* Fridericia's QT correction formula (QTcF) >=450 milliseconds (msec) (if single electrocardiogram [ECG] at screening shows QTcF >=450 msec, a mean of triplicate measurements should be used to confirm that participant meets exclusion criterion).
* Laboratory results as follows

  1. Serum albumin <3.5 grams per deciliter (g/dL)
  2. Glomerular filtration rate (GFR) <60 mL/minute/1.73 per meter square as calculated by the Chronic kidney disease- Epidemiologic Collaboration (CKD-EPI) formula.
  3. International normalized Ratio (INR) >1.25
  4. Platelet count <140 times 10^9/liter (L)
  5. Total bilirubin >1.25 times ULN

     1. For participants with benign unconjugated hyperbilirubinemia with total bilirubin >1.25 times ULN, discussion for inclusion to the study is required with the Medical Monitor
  6. Urine albumin to creatinine ratio (ACR) >=0.03 mg/mg (or >=30 mg/g). In the event of an ACR above this threshold, eligibility may be confirmed by a second measurement 1) In cases where participants have low urine albumin and low urine creatinine levels resulting in a urine ACR calculation >=0.03 mg/mg (or >=30 mg/g), the investigator should confirm that the participant does not have a history of diabetes, hypertension or other risk factors that may affect renal function and discuss with the Medical Monitor, or designee.
* History of/sensitivity to GSK3228836 or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Boston, Massachusetts, United States
- GSK Investigational Site, Toronto, Ontario, Canada
- GSK Investigational Site, Rotterdam, Netherlands
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label, single arm study to mechanistically interrogate the therapeutic effect of GSK3228836 in participants with Chronic Hepatitis B via intrahepatic immunophenotyping.
Pre-assignment Details: A total of 12 participants were enrolled in this study.
Groups:
- GSK3228836 300 mg: Participants on stable nucleos(t)ide therapy received GSK3228836 300 milligrams (mg) administered subcutaneously (SC) weekly once for 12 weeks along with a loading dose of GSK3228836 300 mg in Week 1 (Day 4) and Week 2 (Day 11).
Period: Overall Study
Arm/Group | GSK3228836 300 mg
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.8 (8.48)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender categories (with 0<n<11) are combined into one 'De-identified' category to maintain participant confidentiality and privacy, as they could lead to participant re-identification.
  Participants
    De-identified | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race categories (with 0<n<11) are combined into one 'De-identified' category to maintain participant confidentiality and privacy, as they could lead to participant re-identification.
  Participants
    De-identified | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Serum Hepatitis B Virus Surface Antigen (HBsAg) Level Less Than (<) Lower Limit of Quantitation (LLOQ)
Description: Percentage of participants achieving serum HBsAg level <LLOQ were reported. Percentage values are rounded-off.
Time Frame: Up to Week 12
Population: Intent to Treat (ITT) Set that included all participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 12
Percentage of participants | 25

2. Secondary Outcome: Percentage of Participants With Sustained HBsAg Response (HBsAg <LLOQ) for 24 Weeks After the Planned and Actual End of GSK3228836 Treatment
Description: Sustained HBsAg response is defined as HBsAg <LLOQ for 24 weeks from end of GSK3228836 treatment. Percentage values are rounded-off.
Time Frame: Up to 24 weeks off treatment (Study Weeks 12 to 36)
Population: Intent to Treat (ITT) Set that included all participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 12
Percentage of participants
  Sustained HBsAg Response for 24 Weeks after Planned End of GSK3228836 Treatment | 8
  Sustained HBsAg Response for 24 Weeks after Actual End of GSK3228836 Treatment | 8

3. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response (HBsAg <LLOQ and HBV DNA <LLOQ) for 24 Weeks After the Planned and Actual End of GSK3228836 Treatment
Description: Sustained virologic response is defined as HBsAg <LLOQ and hepatitis B virus (HBV) deoxyribonucleic acid (DNA) <LLOQ for 24 weeks from end of GSK3228836 treatment. Percentage values are rounded-off.
Time Frame: Up to 24 weeks off treatment (Study Weeks 12 to 36)
Population: Intent to Treat (ITT) Set that included all participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 12
Percentage of participants
  Sustained Virologic Response for 24 Weeks after Planned End of GSK3228836 Treatment | 8
  Sustained Virologic Response for 24 Weeks after Actual End of GSK3228836 Treatment | 8

4. Secondary Outcome: Percentage of Participants Achieving HBsAg <LLOQ at Indicated Time Points
Description: Percentage of participants achieving HBsAg <LLOQ were assessed at indicated time points. Percentage values are rounded-off.
Time Frame: Baseline (Week -1), treatment Day 78 and off treatment (OT) Day 162
Population: Intent to Treat (ITT) Set that included all participants who received at least one dose of study treatment. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the 'Overall Number of Participants Analyzed' field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 12
Percentage of participants
  Baseline (Week -1) | 0
  Treatment Day 78: number analyzed (Participants) | 10
  Treatment Day 78 | 30
  Off Treatment Day 162: number analyzed (Participants) | 11
  Off Treatment Day 162 | 18

5. Secondary Outcome: Percentage of Participants Achieving HBV DNA <LLOQ at Indicated Time Points
Description: Percentage of participants achieving HBV DNA <LLOQ were assessed at indicated time points. Percentage values are rounded-off.
Time Frame: Baseline (Week -1), treatment Day 78 and off treatment Day 162
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 12
Percentage of participants
  Baseline (Week -1) | 92
  Treatment Day 78: number analyzed (Participants) | 9
  Treatment Day 78 | 78
  Off Treatment Day 162: number analyzed (Participants) | 11
  Off Treatment Day 162 | 100

6. Secondary Outcome: Percentage of Participants Achieving HBsAg <LLOQ and HBV DNA <LLOQ at Indicated Time Points
Description: Percentage of participants achieving HBsAg <LLOQ and HBV DNA <LLOQ were assessed at indicated time points. Percentage values are rounded-off.
Time Frame: Baseline (Week -1), treatment Day 78 and off treatment Day 162
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 12
Percentage of participants
  Baseline (Week -1) | 0
  Treatment Day 78: number analyzed (Participants) | 10
  Treatment Day 78 | 20
  Off Treatment Day 162: number analyzed (Participants) | 11
  Off Treatment Day 162 | 18

7. Secondary Outcome: Percentage of Participants With Categorical Change From Baseline in HBsAg Values at Indicated Time Points
Description: Participants who achieved a decline in HBsAg values from Baseline were reported. Participants were categorized in the following categorical HBsAg decline of <0.5, greater than or equal to (>=) 0.5, >=1, >=1.5, and >=3 log10 international units per milliliter (IU/mL). The 'HBsAg < LLOQ' category is derived based on Absolute/raw HBsAg result. The HBsAg decline categories are based on change from Baseline values. Percentage values are rounded-off.
Time Frame: Baseline (Week -1), Treatment Week 12 and off treatment Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 11
Percentage of participants
  Treatment Week 12, HBsAg < LLOQ: number analyzed (Participants) | 10
  Treatment Week 12, HBsAg < LLOQ | 30
  Treatment Week 12, HBsAg decline <0.5 log10 IU/mL: number analyzed (Participants) | 10
  Treatment Week 12, HBsAg decline <0.5 log10 IU/mL | 10
  Treatment Week 12, HBsAg decline >=0.5 log10 IU/mL: number analyzed (Participants) | 10
  Treatment Week 12, HBsAg decline >=0.5 log10 IU/mL | 90
  Treatment Week 12, HBsAg decline >=1 log10 IU/mL: number analyzed (Participants) | 10
  Treatment Week 12, HBsAg decline >=1 log10 IU/mL | 80
  Treatment Week 12, HBsAg decline >=1.5 log10 IU/mL: number analyzed (Participants) | 10
  Treatment Week 12, HBsAg decline >=1.5 log10 IU/mL | 80
  Treatment Week 12, HBsAg decline >=3 log10 IU/mL: number analyzed (Participants) | 10
  Treatment Week 12, HBsAg decline >=3 log10 IU/mL | 50
  Off Treatment Week 24, HBsAg < LLOQ | 18
  Off Treatment Week 24, HBsAg decline <0.5 log10 IU/mL | 73
  Off Treatment Week 24, HBsAg decline >=0.5 log10 IU/mL | 27
  Off Treatment Week 24, HBsAg decline >=1 log10 IU/mL | 27
  Off Treatment Week 24, HBsAg decline >=1.5 log10 IU/mL | 27
  Off Treatment Week 24, HBsAg decline >=3 log10 IU/mL | 18

8. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT) Greater Than (>)3 Times Upper Limit of Normal (ULN) at Indicated Time Points
Description: Blood samples were collected at indicated time points to assess ALT levels. The ALT normalization (ALT <=upper limit of normal [ULN]) over time in absence of rescue medication in participants with Baseline ALT>ULN and ALT data at that visit. Participants who achieved ALT normalization were reported.
Time Frame: Baseline (Week -1), treatment Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78; off treatment Days 1, 8, 22, 50, 78, 106, 134 and 162
Population: Intent to Treat (ITT) Set that included all participants who received at least one dose of study treatment. The "n" represents the number of participants with Baseline ALT > ULN and ALT data at that visit. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the 'Overall Number of Participants Analyzed' field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 12
Participants
  Baseline (Week -1) | 0
  Treatment Day 8 | 0
  Treatment Day 15: number analyzed (Participants) | 11
  Treatment Day 15 | 0
  Treatment Day 22 | 0
  Treatment Day 29: number analyzed (Participants) | 11
  Treatment Day 29 | 0
  Treatment Day 36: number analyzed (Participants) | 11
  Treatment Day 36 | 1
  Treatment Day 43: number analyzed (Participants) | 10
  Treatment Day 43 | 1
  Treatment Day 50: number analyzed (Participants) | 10
  Treatment Day 50 | 1
  Treatment Day 57: number analyzed (Participants) | 10
  Treatment Day 57 | 1
  Treatment Day 64: number analyzed (Participants) | 11
  Treatment Day 64 | 1
  Treatment Day 71: number analyzed (Participants) | 11
  Treatment Day 71 | 1
  Treatment Day 78: number analyzed (Participants) | 11
  Treatment Day 78 | 0
  Off Treatment Day 1: number analyzed (Participants) | 10
  Off Treatment Day 1 | 0
  Off Treatment Day 8: number analyzed (Participants) | 11
  Off Treatment Day 8 | 0
  Off Treatment Day 22: number analyzed (Participants) | 11
  Off Treatment Day 22 | 0
  Off Treatment Day 50: number analyzed (Participants) | 11
  Off Treatment Day 50 | 0
  Off Treatment Day 78: number analyzed (Participants) | 9
  Off Treatment Day 78 | 0
  Off Treatment Day 106: number analyzed (Participants) | 11
  Off Treatment Day 106 | 1
  Off Treatment Day 134: number analyzed (Participants) | 9
  Off Treatment Day 134 | 0
  Off Treatment Day 162: number analyzed (Participants) | 11
  Off Treatment Day 162 | 0

9. Secondary Outcome: Number of Participants With HBe Antibody (Anti-HBeAg) Levels
Description: Blood samples were collected to assess HBe antibody levels and results reported are for Baseline HBeAg positive participants.
Time Frame: Baseline (Week -1), treatment Days 29, 36, and 57; off treatment Days 1, 8, 22, 50, 78, 106, 134 and 162
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 12
Participants
  Baseline (Week -1) | 11
  Treatment Day 29: number analyzed (Participants) | 11
  Treatment Day 29 | 11
  Treatment Day 36: number analyzed (Participants) | 1
  Treatment Day 36 | 0
  Treatment Day 57: number analyzed (Participants) | 10
  Treatment Day 57 | 9
  Off Treatment Day 1: number analyzed (Participants) | 10
  Off Treatment Day 1 | 9
  Off Treatment Day 8: number analyzed (Participants) | 11
  Off Treatment Day 8 | 10
  Off Treatment Day 22: number analyzed (Participants) | 11
  Off Treatment Day 22 | 10
  Off Treatment Day 50: number analyzed (Participants) | 11
  Off Treatment Day 50 | 10
  Off Treatment Day 78: number analyzed (Participants) | 11
  Off Treatment Day 78 | 10
  Off Treatment Day 106: number analyzed (Participants) | 11
  Off Treatment Day 106 | 10
  Off Treatment Day 134: number analyzed (Participants) | 9
  Off Treatment Day 134 | 8
  Off Treatment Day 162: number analyzed (Participants) | 11
  Off Treatment Day 162 | 10

10. Secondary Outcome: Actual Values of HBsAg at Indicated Time Points
Description: Blood samples were collected from participants at indicated time points to assess HBsAg levels.
Time Frame: Baseline (Week -1), treatment Day 78 and off treatment Day 162
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 12
Log10 IU/mL
  Baseline (Week -1) | 3.29 (0.590)
  Treatment Day 78: number analyzed (Participants) | 10
  Treatment Day 78 | 0.33 (1.432)
  Off Treatment Day 162: number analyzed (Participants) | 11
  Off Treatment Day 162 | 2.08 (1.933)

11. Secondary Outcome: Mean Change From Baseline in HBsAg at Indicated Time Points
Description: Blood samples were collected from participants at indicated time points to assess HBsAg levels. Change from Baseline was defined as value at the indicated time point minus Baseline value. Baseline was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Week -1), treatment Day 78 and off treatment Day 162
Population: Intent to Treat (ITT) Set that included all participants who received at least one dose of study treatment. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the 'Overall Number of Participants Analyzed' field. 'Number Analyzed' signifies participants evaluable for the specified time points. Participants who had Baseline and at least 1 post-Baseline visit values were included in analysis.
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 11
Log10 IU/mL
  Treatment Day 78: number analyzed (Participants) | 10
  Treatment Day 78 | -2.923 (1.5803)
  Off Treatment Day 162 | -1.183 (1.8343)

12. Secondary Outcome: Actual Values of HBV DNA at Indicated Time Points
Description: Blood samples were collected from participants at indicated time points to assess HBV DNA levels.
Time Frame: Baseline (Week -1), treatment Day 78 and off treatment Day 162
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 12
Log10 IU/mL
  Baseline (Week -1) | 0.43 (0.849)
  Treatment Day 78: number analyzed (Participants) | 9
  Treatment Day 78 | 0.31 (0.611)
  Off Treatment Day 162: number analyzed (Participants) | 11
  Off Treatment Day 162 | 0.24 (0.525)

13. Secondary Outcome: Mean Change From Baseline in HBV DNA at Indicated Time Points
Description: Blood samples were collected from participants at indicated time points to assess HBV DNA levels. Change from Baseline was defined as value at the indicated time point minus Baseline value. Baseline was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Week -1), treatment Day 78 and off treatment Day 162
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 11
Log10 IU/mL
  Treatment Day 78: number analyzed (Participants) | 9
  Treatment Day 78 | -0.271 (1.1145)
  Off Treatment Day 162 | -0.237 (0.7871)

14. Secondary Outcome: Actual Values of HB Surface Antibody (Anti-HBsAg) Levels at Indicated Time Points
Description: Blood samples were collected from participants at indicated time points to assess anti-HBsAg levels.
Time Frame: Baseline (Week -1) and off treatment Days 1 and 162
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 12
Log10 IU/mL
  Baseline (Week -1) | 0.60 (0.000)
  Off Treatment Day 1: number analyzed (Participants) | 10
  Off Treatment Day 1 | 0.71 (0.238)
  Off Treatment Day 162: number analyzed (Participants) | 11
  Off Treatment Day 162 | 0.70 (0.260)

15. Secondary Outcome: Area Under the Concentration-time Curve (AUC) for ALT at Indicated Time Points
Description: Blood samples were collected from participants to assess AUC for ALT. On-treatment blood samples were collected from Weeks 1 to 12 and follow-up blood samples were collected from Weeks 12 to 36. AUC was calculated and presented for on-treatment (12 Weeks), follow-up (24 weeks), and On-treatment + follow-up (Weeks 1 to 36).
Time Frame: Study Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 16, 20, 24, 28, 32 and 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Weeks*International Units Per Liter
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 12
Weeks*International Units Per Liter
  On-Treatment (12 Weeks) | 494.75 (562.593)
  Follow-up (24 weeks): number analyzed (Participants) | 11
  Follow-up (24 weeks) | 650.58 (462.762)
  On-Treatment + Follow-Up (Weeks 1 to 36): number analyzed (Participants) | 11
  On-Treatment + Follow-Up (Weeks 1 to 36) | 1173.72 (836.768)

16. Secondary Outcome: Time to Maximum ALT
Description: Time to maximum ALT (maximum peak in ALT) during 36 week (treatment + follow-up) is defined as time from Baseline to the time of first peak in ALT.
Time Frame: Up to Study Week 36
Population: Intent to Treat (ITT) Set that included all participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | GSK3228836 300 mg
Number analyzed (Participants) | 12
Weeks | NA [27.1 to NA] — NA indicates median and 95% CI (upper limit) could not be derived, as <50% of participants experienced the event within the treatment arm.

ADVERSE EVENTS:
Time Frame: Up to Study Week 36
Description: All-cause mortality, Serious adverse events and non-serious adverse events were reported for the Safety Population which consisted of all participants who received at least one dose of study treatment.
Arm/Group | GSK3228836 300 mg
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3228836 300 mg (N=12)
Injection site erythema (General disorders) | 7 (30)
Injection site pruritus (General disorders) | 4 (18)
Fatigue (General disorders) | 2 (2)
Injection site bruising (General disorders) | 2 (10)
Injection site pain (General disorders) | 2 (40)
Pyrexia (General disorders) | 2 (2)
Chest discomfort (General disorders) | 1 (1)
Injection site discomfort (General disorders) | 1 (1)
Injection site swelling (General disorders) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Sensory disturbance (Nervous system disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT04544956/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT04544956/SAP_001.pdf